CLINICAL TRIAL: NCT06948058
Title: Clinical Research Evaluating Smoking Cessation With E-Cigarettes and Nicotine Therapy
Acronym: CRESCENT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00000326; P20GM130414 (NIH)
Record Dates: First submitted 2025-04-22; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Smoking Cessation; Obesity and Obesity-related Medical Conditions
Keywords: obesity; electronic cigarettes; harm reduction
MeSH Terms: conditions — Smoking Cessation; Obesity; Vaping; Harm Reduction | interventions — Electronic Nicotine Delivery Systems; Nicotine Replacement Therapy

STUDY DESIGN:
Intervention Model Description: A 3-group design.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor will not know the outcome of randomized assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Electronic Cigarette (EC) Condition (Experimental): Participants in this condition will receive the EC intervention.
  Interventions: Other: Electronic Cigarettes (EC)
- Nicotine Replacement Therapy Condition (Experimental): Participants in this condition will receive the NRT intervention.
  Interventions: Other: Nicotine replacement therapy (NRT)
- No-Product Control Condition (CON) (No Intervention): Participants in this condition will not receive any alternate nicotine product.

INTERVENTIONS:
Other: Electronic Cigarettes (EC) — Participants will receive information about the comparative risk of alternative nicotine products relative to smoking and will be asked to switch to EC for 8 weeks, with EC provided.
  Arms: Electronic Cigarette (EC) Condition
Other: Nicotine replacement therapy (NRT) — Participants will receive information about the comparative risk of alternative nicotine products relative to smoking and will be asked to switch to combination NRT (transdermal + oral) for 8 weeks, with NRT provided.
  Arms: Nicotine Replacement Therapy Condition

SUMMARY:
This project will investigate the effects of alternative nicotine products on smoking, weight gain, and related outcomes.

DETAILED DESCRIPTION:
The purpose of this study is to provide preliminary information on the effect of electronic cigarettes (EC) and nicotine replacement therapy (NRT) among SWO. This study will randomize up to 60 individuals who smoke cigarettes with comorbid obesity (SWO) to receive (1) electronic cigarettes (EC), (2) nicotine replacement therapy (NRT), or 3) a no-product control (CON) condition for 8 weeks. Assessments will occur at baseline, and 1, 2, and 3-months follow-up, aiming: 1) To compare EC, NRT, and CON on smoking, exhaled carbon monoxide, and number of quit attempts; 2) To compare EC and NRT on acceptability and adherence; 3) To compare EC, NRT, and CON effects on weight, central adiposity, glucose regulation, inflammation, cotinine, and blood pressure at follow-up.

ELIGIBILITY:
Inclusion Criteria:

* body mass index (BMI) ≥ 30 kg/m2 (i.e., obese)
* smoked ≥ 5 cigarettes/day during the past year
* 21 or older (due to minimum legal age EC restrictions)
* exhaled breath carbon monoxide (CO) level > 6 ppm at Baseline (BL) (to confirm self-reported smoking)
* willing to use EC or NRT for 8 weeks
* access to a Bluetooth-enabled smartphone/tablet (to permit remote measurement of CO and other outcome variables)

Exclusion Criteria:

* received smoking cessation treatment of any kind in the past 30 days (actively quitting smoking),
* currently using EC or NRT more than 2 days/week (this may affect responses to study-supplied products)
* hospitalized for mental illness in past 30 days
* heart-related event (e.g., heart attack, severe angina) in past 30 days
* residing with another person currently enrolled in the study
* pregnant, nursing, or planning to become pregnant in the next 6 months
* medical contraindication for study or product use (e.g., allergy to adhesives)
* taken prescription weight loss medication in the last 30 days

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
number of cigarettes per day | 2 months
  Daily use of cigarettes will be determined using the Timeline Follow-Back (TLFB) in follow-up assessments.
carbon monoxide (CO) | 2 months
  Exhaled breath sample used to measure carbon monoxide
number of quit attempts | 2 months
  Number of attempts to quit smoking during the experimental period

SECONDARY OUTCOMES:
product acceptability | 2 months
  Self-rated acceptability (e.g., satisfaction) of the alternative nicotine product assigned (if applicable)
product adherence | 2 months
  Percentage of days using the alternative nicotine product assigned (if applicable)
change in weight | 2 months
  change in body weight (lbs) from baseline to 2 months
change in waist circumference | 2 months
  change in waist circumference, a measure of central adiposity, from baseline to 2 months
A1c | 2 months
  level of A1c, measured via blood sample, as a measure of glucose regulation
interleukin-6 (IL-6) | 2 months
  level of IL-6, measured via blood sample, as a measure of inflammation
cotinine | 2 months
  level of cotinine, measured via blood sample, as a measure of nicotine exposure
diastolic blood pressure | 2 months
  diastolic blood pressure measured using a cuff
systolic blood pressure | 2 months
  systolic blood pressure measured using a cuff

CONTACTS AND LOCATIONS:
Locations (1):
- Brown University, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be kept and used for future research on chronic disease and substance use.
Time Frame: Clinical Laboratory Core data collected to fulfill the aims of the Center for Addiction and Disease Risk Exacerbation will be available to request immediately following publication, with no prespecified end date.
Access Criteria: After all data are collected and the results of the study are published, deidentified data and biospecimens may be made available to other qualified investigators at Brown or other institutions upon request. The request will be evaluated by the investigators to ensure that it meets reasonable demands of scientific integrity.